CLINICAL TRIAL: NCT01897415
Title: Phase I Clinical Trial of Autologous Mesothelin Re-directed T Cells in Patients With Chemotherapy Refractory Metastatic Pancreatic Cancer
Brief Title: Autologous Redirected RNA Meso CAR T Cells for Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08212
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Subjects With Metastatic Pancreatic Ductal Adenocarcinoma (PDA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous T cells (Experimental): Autologous T cells transfected with chimeric anti-mesothelin immunoreceptor SS1
  Interventions: Biological: Autologous T cells transfected with chimeric anti-mesothelin immunoreceptor SS1

INTERVENTIONS:
Biological: Autologous T cells transfected with chimeric anti-mesothelin immunoreceptor SS1

SUMMARY:
This is a Phase I safety and feasibility study. Subjects will be enrolled serially. For subject safety, the preceding subject must have completed one cycle of therapy (28 days) before the next subject can be treated. Subjects will be treated with i.v. administration of 1 to 3e8 per meter squared RNA CAR T cells three times weekly (M-W-F) for three weeks.

DETAILED DESCRIPTION:
This phase I study is being conducted to establish safety and feasibility of intravenous (IV) RNA mesothelin re-directed autologous T cell administration in patients with chemotherapy-refractory metastatic pancreatic cancer.

Subjects will be enrolled serially. For subject safety, the preceding subject must have completed therapy and be 28 days from their last infusion before the next subject can be treated.. Subjects will be treated with IV administration of 1 to 3e8/m2 RNA CAR T cells three times weekly (M-W-F) for three weeks.

Main eligibility criteria: Subjects with metastatic pancreatic ductal adenocarcinoma (PDA) who have chemotherapy-refractory disease. Inclusion criteria include patients older than 18 years of age diagnosed with metastatic PDA with ECOG 0-1 performance status and 3 month expected survival. Exclusion criteria include a pericardial effusion, active autoimmune disease requiring immunosuppressive therapy, active anti-coagulation therapy, known HIV or HTLV I/II positivity, prior treatment with murine monoclonal antibodies or history of allergy to murine proteins.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic pancreatic adenocarcinoma.
* Patients greater than or equal to 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy greater than 3 months.
* Evidence of metastatic disease and failure of at least 1 prior chemotherapy for metastatic disease.
* Subjects must have measureable disease as defined by RECIST 1.1 criteria.
* Satisfactory organ and bone marrow function
* Blood coagulation parameters: PT such that international normalized ratio (INR) is less than or equal to 1.5 (or an in-range INR, usually between 2 and 3, if a subject is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thromboembolus) and a PTT less than or equal to 1.2 time the upper limit of normal.
* Subjects must have adequate venous peripheral access for apheresis. Patients must also have adequate venous access for subsequent modified CAR T cell administration which can be done through a central venous access (e.g. port for systemic chemotherapy)
* Ability to understand and the willingness to provide written informed consent.
* Short-term therapy for acute conditions not specifically related to pancreatic cancer is allowed if such therapy does not include immune modulating agents.
* Male and Female subjects agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) during the study and for 3 months following the last dose of the study cell infusion.
* Subject must understand and sign the study-specific informed consent.

Exclusion Criteria:

* Participated in any other trial in which receipt of an investigational study drug occurred within 28 days (42 days for non-murine monoclonal antibodies) prior to entry into the study.
* Received any anticancer medication in the 2 weeks (i.e. 14 days) prior to receiving their first dose of study treatment and no other concurrent chemotherapy or immunotherapy (e.g. monoclonal antibodies)
* Active invasive cancer other than pancreatic adenocarcinoma. Patients with active non-invasive cancers (such as non-melanoma skin cancer, superficial cervical and bladder and prostate cancer with PSA level less than 1.0) are not excluded.
* Known HIV, HCV, and HBV positive
* Active autoimmune disease (including but not limited to: systemic lupus erythromatosis, Sjogrens syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) requiring immunosuppressive therapy within the past 4 weeks, with exception of thyroid replacement.
* Patients with ongoing or active infection.
* Planned concurrent treatment with systemic high dose corticosteroids.
* Prior gene therapy or therapy with murine monoclonal antibodies or products of murine origin.
* Concurrent treatment with any anticancer agent.
* History of allergy to murine proteins
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
* Any clinically significant pericardial effusion; CHF (NY Heart Association Grade II-IV) or cardiovascular condition that would preclude assessment of mesothelin induced pericarditis.
* Subjects on active anti-coagulation therapy.
* Pregnant women are excluded from this study because autologous transduced T cells may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants, secondary to treatment of the mother with autologous transduced T cells, breastfeeding should be discontinued if the mother is treated.
* Feasibility assessment demonstrates less than 20% transfection of target lymphocytes or insufficient expansion of modified CAR T cells to complete 9 infusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Beatty, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States